CLINICAL TRIAL: NCT05955521
Title: Development of a Prognostic and Predictive Biomarker for Locally Advanced Breast Cancer Patients Treated With Neoadjuvant Chemotherapy Using Exosome
Brief Title: Exosome as the Prognostic and Predictive Biomarker in EBC Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JI-YEON, KIM, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EXO_Breast
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Triple Negative Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CtDNA/Exosome evaluation (Experimental)
  Interventions: Procedure: exosome and ctDNA evaluation

INTERVENTIONS:
Procedure: exosome and ctDNA evaluation — Serial exosome and ctDNA evaluation during follow up period between neoadjuvant chemotherapy and surveillance after curative surgery.

SUMMARY:
This study is the experimental study for serial ctDNA and exosome evaluation in EBC patients

ELIGIBILITY:
Inclusion Criteria:

* Early breast cancer
* Planned neoadjuvant chemotherapy
* Triple negative breast cancer or HER2-positive breast cancer

Exclusion Criteria:

* Stage IV breast cancer
* Hormone receptor positive breast cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Prognostic biomarker for EBC | 60 months
  Positive predictive value of ctDNA/Exosome for BC recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Ji-Yeon Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No